CLINICAL TRIAL: NCT06139601
Title: A Single Session Community-Based Body Empowerment Session
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Equip Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EH1006
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Body Image
Keywords: body image; eating disorder; psychological wellbeing; weight stigma; social stigma; digital health
MeSH Terms: conditions — Feeding and Eating Disorders; Weight Prejudice; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Body empowerment intervention program (Other): All study participants will complete a single session body empowerment program.
  Interventions: Behavioral: Virtual single session intervention

INTERVENTIONS:
Behavioral: Virtual single session intervention — A single session, self-paced body empowerment program. The program consists of a single 45-minute self paced, interactive, virtual module.

SUMMARY:
This present study will examine the effectiveness of a single session, virtually delivered body empowerment program for decreasing participants thin ideal internalization. The intervention asks participants to identify cultural norms surrounding appearance and attractiveness, then challenge these ideals. Participants will answer questions about thin ideal internalization before and after the program.

DETAILED DESCRIPTION:
A body empowerment program rooted in the psychological theory of cognitive dissonance has been shown to be effective to reduce the value of the thin beauty ideal. This theory proposes that humans are motivated to maintain consistency in their beliefs and actions, and inconsistencies will result in psychological discomfort (or cognitive dissonance). A shift in beliefs or actions is required to resolve this discomfort and maintain consistency. However, the accessibility of this program is lacking. The proposed study will examine the effectiveness of a single session, virtually delivered body empowerment program designed to create cognitive dissonance by asking participants to identify cultural norms surrounding appearance and attractiveness, then challenge these ideals through a series of interactive activities in a fully virtual, self-paced module. Challenging these ideals (e.g., identifying how ideals represent very narrow identities and are informed by oppressive value systems, stating the psychological costs of trying to change your body to match ideals) theoretically creates cognitive dissonance in those who have internalized the value of pursuing those ideals. This dissonance is resolved through a reduced investment in the ideals and then hypothesized to lead to more positive attitudes about body image, dieting, and other unhealthy weight control behaviors. The program consists of a single 45-minute self paced, interactive, virtual module. Primary assessments will be completed at pre-intervention and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Able to reliably access internet
* Can speak and read English
* Completed the body empowerment program

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in thin ideal internalization | Pre intervention obtained prior to completing the intervention, and immediately following the intervention.
  Sociocultural Attitudes Towards Appearance Questionnaire (SATAQ-4) questionnaire will be used to evaluate thin ideal internalization. Participants note their agreement or disagreement regarding beliefs about appearance on a 5-point Likert scale ranging from definitely disagree (1) to definitely agree (5). The thin ideal internalization subscale will be used. High scores indicate greater thin ideal internalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Equip Health, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghaderi A, Stice E, Andersson G, Eno Persson J, Allzen E. A randomized controlled trial of the effectiveness of virtually delivered Body Project (vBP) groups to prevent eating disorders. J Consult Clin Psychol. 2020 Jul;88(7):643-656. doi: 10.1037/ccp0000506. PMID 32551736
- [Background] Butryn ML, Rohde P, Marti CN, Stice E. Do participant, facilitator, or group factors moderate effectiveness of the Body Project? Implications for dissemination. Behav Res Ther. 2014 Oct;61:142-9. doi: 10.1016/j.brat.2014.08.004. Epub 2014 Aug 20. PMID 25199580
- [Background] Stice E, Rohde P, Shaw H, Gau JM. Clinician-led, peer-led, and internet-delivered dissonance-based eating disorder prevention programs: Acute effectiveness of these delivery modalities. J Consult Clin Psychol. 2017 Sep;85(9):883-895. doi: 10.1037/ccp0000211. Epub 2017 Apr 20. PMID 28425735
- [Background] Stice E, Bohon C, Shaw H, Desjardins CD. Efficacy of virtual delivery of a dissonance-based eating disorder prevention program and evaluation of a donation model to support sustained implementation. J Consult Clin Psychol. 2023 Mar;91(3):139-149. doi: 10.1037/ccp0000796. Epub 2023 Feb 6. PMID 36745074
- [Background] Stice E, Marti CN, Shaw H, Rohde P. Meta-analytic review of dissonance-based eating disorder prevention programs: Intervention, participant, and facilitator features that predict larger effects. Clin Psychol Rev. 2019 Jun;70:91-107. doi: 10.1016/j.cpr.2019.04.004. Epub 2019 Apr 8. PMID 31004832
- [Background] Freijy T, Kothe EJ. Dissonance-based interventions for health behaviour change: a systematic review. Br J Health Psychol. 2013 May;18(2):310-37. doi: 10.1111/bjhp.12035. PMID 23480429
- [Background] Schleider JL, Dobias ML, Sung JY, Mullarkey MC. Future Directions in Single-Session Youth Mental Health Interventions. J Clin Child Adolesc Psychol. 2020 Mar-Apr;49(2):264-278. doi: 10.1080/15374416.2019.1683852. Epub 2019 Dec 4. PMID 31799863
- [Background] Schleider JL, Weisz JR. Little Treatments, Promising Effects? Meta-Analysis of Single-Session Interventions for Youth Psychiatric Problems. J Am Acad Child Adolesc Psychiatry. 2017 Feb;56(2):107-115. doi: 10.1016/j.jaac.2016.11.007. Epub 2016 Nov 25. PMID 28117056